CLINICAL TRIAL: NCT02540239
Title: Premedication Simethione Improves Visibility During Bowel Cleansing for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Tongji Hospital (Other); Qilu Hospital of Shandong University (Other); Zhongda Hospital (Other); Jinan Military General Hospital (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, fangjun, Digestive Endoscopy Center, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: simethione
Record Dates: First submitted 2015-03-02; First posted 2015-09-03 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Bowel Preparation Scale; the Amount of Air Bubble; Adenoma Detection Rate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2L PEG (Placebo Comparator): only used 2L PEG
  Interventions: Drug: 2L PEG
- Simethione+2L PEG (Experimental): used 2L PEG+Simethione
  Interventions: Drug: 2L PEG+simethicone

INTERVENTIONS:
Drug: 2L PEG
  Arms: 2L PEG
Drug: 2L PEG+simethicone
  Arms: Simethione+2L PEG

SUMMARY:
To evaluate the efficacy, visibility of low volume polyethyleneglycol-simeticone (2-LPEG-S) for colonoscopy.

DETAILED DESCRIPTION:
In this randomized controlled study, consecutive outpatients scheduled for elective colonoscopy were randomized into two groups. Group A patients (n = 300) used only 2 L PEG before colonoscopy. Patients in group B (n = 300) were additionally advised to simeticone plus 2 L PEG, The overall quality of colonoscopy cleaning was evaluated using the Boston Bowel Preparation Scale by a single endoscopist who was blinded to the intervention. Visibility was blindly assessed for the amount of air bubbles and adenoma detection rate (ADR). Difficulty of procedure, and adverse events were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients are between 18-65 years old
* undergoing colonoscopy for diagnostic investigation, colorectal cancer screening or follow-up

Exclusion Criteria:

* suspected gastrointestinal obstruction or perforation
* severe acute inflammatory bowel disease
* toxic megacolon
* ileus or gastric retention, ileostomy,
* hypersensitivity to any of the ingredients
* pregnancy and lactation and/or at a risk of becoming pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | 2 days
bowel preparation scale | 2 days
the amount of air bubbles | 2 days
  Five areas of the colon (rectosigmoid, descending, transverse, ascending, and cecum) were graded for the amount of air bubbles.The amount of intraluminal air bubbles was classified into four grades as shown below: Grade 0 = No or minimal scattered bubbles; Grade 1 = Bubbles covering at least half the luminal diameter; Grade 2 = Bubbles covering the circumference of the lumen; Grade 3 = Bubbles filling the entire lumen.

CONTACTS AND LOCATIONS:
Overall Officials: LI ZHAO SHEN, M.D, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Di Nardo G, Aloi M, Cucchiara S, Spada C, Hassan C, Civitelli F, Nuti F, Ziparo C, Pession A, Lima M, La Torre G, Oliva S. Bowel preparations for colonoscopy: an RCT. Pediatrics. 2014 Aug;134(2):249-56. doi: 10.1542/peds.2014-0131. Epub 2014 Jul 7. PMID 25002661
- [Background] Gentile M, De Rosa M, Cestaro G, Forestieri P. 2 L PEG plus ascorbic acid versus 4 L PEG plus simethicon for colonoscopy preparation: a randomized single-blind clinical trial. Surg Laparosc Endosc Percutan Tech. 2013 Jun;23(3):276-80. doi: 10.1097/SLE.0b013e31828e389d. PMID 23751992
- [Derived] Bai Y, Fang J, Zhao SB, Wang D, Li YQ, Shi RH, Sun ZQ, Sun MJ, Ji F, Si JM, Li ZS. Impact of preprocedure simethicone on adenoma detection rate during colonoscopy: a multicenter, endoscopist-blinded randomized controlled trial. Endoscopy. 2018 Feb;50(2):128-136. doi: 10.1055/s-0043-119213. Epub 2017 Oct 6. PMID 28985630